CLINICAL TRIAL: NCT01057628
Title: Phase III Study of ASP1941 -A Phase III, Randomized, Double-Blind, Placebo-controlled, Monotherapy Study to Assess the Efficacy, Safety, and Tolerability of ASP1941 in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess the Efficacy and Safety of ASP1941 in Japanese Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0105
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Blood glucose; ASP1941; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1941 group (Experimental): oral
  Interventions: Drug: ipragliflozin
- placebo group (Placebo Comparator): oral
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ipragliflozin — oral
  Other Names: ASP1941
  Arms: ASP1941 group
Drug: placebo — oral
  Arms: placebo group

SUMMARY:
This study is to compare the efficacy and safety of ASP1941 with placebo in Japanese patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients for at least 12 weeks
* HbA1c value between 7.0 and 10.0%
* Body Mass Index (BMI) 20.0 - 45.0 kg/m2
* Investigator adjudicates that a subject is able to discontinue currently taking hypoglycemic agents safely during treatment

Exclusion Criteria:

* Type 1 diabetes mellitus patients
* Serum creatinine > upper limit of normal
* Proteinuria (albumin/creatinine ratio > 300mg/g)
* Dysuria and/or urinary tract infection, genital infection
* Significant renal, hepatic or cardiovascular diseases
* Severe gastrointestinal diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-01-13 (Actual); Primary Completion 2010-11-06 (Actual); Study Completion 2010-11-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in HbA1c | 16 weeks

SECONDARY OUTCOMES:
change from baseline in fasting plasma glucose | 16 weeks
change from baseline in fasting serum insulin | 16 weeks
safety as reflected by adverse events, routine safety laboratories, vital signs, physical examinations and 12-lead electrocardiograms (ECGs) | During treatment

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- See also: Link to results on Astellas Clinical Study Results Web site — https://astellasclinicalstudyresults.com/study.aspx?ID=99